CLINICAL TRIAL: NCT04061512
Title: Randomised Phase II/III Study of Rituximab and Ibrutinib (RI) Versus Dexamethasone, Rituximab and Cyclophosphamide (DRC) as Initial Therapy for Waldenström's Macroglobulinaemia
Brief Title: Rituximab and Ibrutinib (RI) Versus Dexamethasone, Rituximab and Cyclophosphamide (DRC) as Initial Therapy for Waldenström's Macroglobulinaemia
Acronym: RAINBOW
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/18/0438
Record Dates: First submitted 2019-07-01; First posted 2019-08-19 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Dexamethasone; Cyclophosphamide; Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DRC Arm (Active Comparator): The DRC arm (chemotherapy) is the control arm and consists of rituximab, cyclophosphamide and dexamethasone. It is widely recommended by international consensus as appropriate treatment for first-line therapy for WM.
  Interventions: Drug: Dexamethasone, cyclophosphamide, rituximab
- RI Arm (Experimental): The RI arm (chemotherapy free) arm will be using the drug ibrutinib, which in combination with rituximab (RI) will be the experimental arm.
  Interventions: Drug: Rituximab, ibrutinib

INTERVENTIONS:
Drug: Dexamethasone, cyclophosphamide, rituximab — DRC Arm (chemotherapy) consists of dexamethasone, cyclophosphamide and rituximab treatment
  Arms: DRC Arm
Drug: Rituximab, ibrutinib — RI Arm (chemotherapy free) consists of rituximab and ibrutinib treatment
  Arms: RI Arm

SUMMARY:
Waldenström's macroglobulinaemia (WM) is a rare type of slow growing lymphoma. It develops when white blood cells grow abnormally.

Typically a disease of the elderly, the median age of presentation is >70 years and the current treatment for WM is unsatisfactory, with incomplete responses and inevitable recurrence. Therefore there is a need to find alternative treatments that are more effective, leading to lasting responses and improved quality of life.

The RAINBOW study is a phase 2-3 trial assessing 'chemotherapy free' treatment as primary therapy for WM which can potentially improve response outcome, durability and importantly, reduce toxicity for WM patients. This approach will be done using the drug Ibrutinib, which in combination with rituximab (RI) will be the experimental arm. As there is no agreed standard on first-line therapy for WM, the control arm is the current treatment based on the most recently published clinical trial results. The control arm consists of rituximab, cyclophosphamide and dexamethasone (DCR), and is widely recommended by international consensus as appropriate treatment for first-line therapy for WM.

In this study, 148 adults (aged ≥ 18 years) with treatment naïve WM will be randomised on a 1:1 ratio to either the treatment or control arm.

Randomised treatment lasts for a maximum of 6 cycles and response will be assessed following 3 cycles of treatment and completion of randomised treatment at approximately 24 weeks after commencing treatment. RI patients may then have up to 5 years of Ibrutinib monotherapy.

Patients will be seen regularly during treatment and then every 3 months for 5 years after treatment discontinuation. Patients will enter annual follow up for survival until the end of trial (including progressed patients).

The study will be conducted at NHS hospitals and is expected to last 9 years and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. Confirmed diagnosis of WM (according to consensus panel / WHO criteria) with measurable IgM paraprotein
3. Previously untreated disease at any stage requiring therapy at the discretion of the treating physician. Suggested criteria for initiating treatment include:

   * haematological suppression to Hb <10g/dl, or neutrophils <1.5x109/l or platelets <150x109/l
   * clinical evidence of hyperviscosity
   * bulky lymphadenopathy and/or bulky splenomegaly
   * presence of B symptoms
4. No previous chemotherapy (prior plasma exchange and steroids are permissible)
5. Eastern Cooperative Oncology Group (ECOG) performance status grade 0 - 2
6. Life expectancy of greater than 6 months
7. Written informed consent
8. Willing to comply with the contraceptive requirements of the trial
9. Negative serum or urine pregnancy test for women of childbearing potential (WOCBP)

Exclusion Criteria:

1. Prior therapy for WM
2. Lymphoplasmacytic lymphoma with no detectable serum IgM paraprotein
3. CNS involvement with WM
4. Autoimmune cytopenias
5. Major surgery within 4 weeks prior to randomisation
6. Clinically significant cardiac disease including the following:

   * Myocardial infarction within 6 months prior to randomisation
   * Unstable angina within 3 months prior to randomisation
   * New York Heart Association class III or IV congestive heart failure
   * History of clinically significant arrhythmias (e.g. sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes)
   * QTcF > 480 msecs based on Fredericia's formula or Bazette's formula
   * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
   * Uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mm Hg
   * Cardiac event within 6 months of screening (e.g. coronary artery stent) requiring dual antiplatelet treatment
7. History of stroke or intracranial haemorrhage within 6 months prior to randomisation
8. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (direct oral anticoagulants (DOACs) allowed)
9. History of severe bleeding disorders considered not to be disease related (Haemophilia A, B or von Willebrand's disease)
10. Requires ongoing treatment with a strong CYP3A inhibitor or inducer
11. Known infection with HIV, or serologic status reflecting active hepatitis B or C infection as follows:

    * Presence of hepatitis B surface antigen (HBsAg). In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive the patient will be excluded
    * Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable
12. Women who are pregnant or breastfeeding or males expecting to conceive or father children at any point from the start of treatment until the end of the "at risk period"
13. Renal failure (creatinine clearance <30 ml/min as estimated by the Cockroft-Gault equation)
14. Patients with chronic liver disease with hepatic impairment Child-Pugh class B or C
15. Known history of anaphylaxis following exposure to rat or mouse derived CDR-grafted humanised monoclonal antibodies.
16. Inability to swallow oral medication
17. Disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (e.g. malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease)
18. Active systemic infection requiring treatment
19. Concomitant treatment with another investigational agent
20. Any life-threatening illness, medical condition, organ system dysfunction, need for profound anticoagulation, or bleeding disorder, which, in the investigator's opinion, could compromise the patient's safety, or put the study at risk
21. Unwilling or unable to take PCP prophylaxis (e.g. cotrimoxazole)
22. History of prior malignancy, with the exception of the following:

    * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to screening and felt to be at low risk for recurrence by treating physician
    * Adequately treated non-melanomatous skin cancer or lentigo maligna melanoma, superficial bladder cancer, carcinoma in situ of the cervix or breast or localized Gleason score 6 prostate cancer without current evidence of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving a preliminary efficacy (response) of the 'chemotherapy free' combination of rituximab and ibrutinib (RI) as primary therapy for WM. | Overall response rate at week 24
Progression free survival (PFS) analysis of rituximab/ibrutinib (RI) when compared to dexamethasone/rituximab/cyclophosphamide (DRC) at 2 years after the last randomisation | 2 years after the last randomisation

SECONDARY OUTCOMES:
Safety and tolerability of RI compared to DRC assessed by the frequency of serious and non-serious adverse events according to CTCAE v5.0 | until 30 calendar days post last IMP administration
Overall response rate (defined as complete response [CR], very good partial response [VGPR], partial response [PR] and minor response [MR]) of RI compared to DRC (at end of randomised treatment and best response over any time point) | through study completion, an average of 2 years.
Time to next treatment | through study completion, an average of 2 years.
Duration of response of RI compared to DRC | through study completion, an average of 2 years.
  (responding patients only)
Overall survival (OS) of patients treated with RI compared to DRC | date of randomisation until the date of death (of any cause)
Quality of Life:EQ-5D-5L questionnaire | 1 year and 2 years after completion of randomised treatment against the baseline quality of life score
  Change in quality of life (QoL) responses in each arm assessed by EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Locations (25):
- United Kingdom (25):
  - Royal United Hospital, Bath, Bath
  - The Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - University Hospital of Wales, Cardiff
  - Colchester Hospital, Colchester
  - Mid Yorkshire NHS Trust, Dewsbury
  - Royal Devon University Hospital, Exeter
  - Medway Maritime Hospital, Gillingham
  - Castle Hill Hospital, Hull
  - NHS Lanarkshire, Lanark
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Barking, Havering and Redbridge University Hospitals NHS Trust, London
  - Barts Health NHS Trust, London
  - King's College Hospital, London
  - Northwick Park Hospital, London
  - University College London Hospitals NHS Foundation Trust, London
  - Christie NHS Foundation Trust, Manchester
  - Norfolk and Norwich Hospital, Norwich
  - Oxford University Hospital, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth
  - Salisbury NHS Foundation Trust, Salisbury
  - Torbay & Newton Abbot Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Hampshire Hospitals NHS Foundation Trust, Winchester

IPD SHARING:
Plan to Share IPD: No